CLINICAL TRIAL: NCT07075406
Title: Real-world Utilization Patterns, Clinical Outcomes, and HCRU in Lower-risk MDS Patients Treated With Luspatercept: A Multinational Medical Record Review Study
Brief Title: A Study to Evaluate Treatment Patterns, Outcomes, and Healthcare Resource Utilization in Patients With Lower-Risk Myelodysplastic Syndromes Treated With Luspatercept
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1043
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Myelodysplastic Syndromes
Keywords: Lower-risk myelodysplastic syndromes (LR-MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants receiving luspatercept treatment
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — According to product label

SUMMARY:
The purpose of this study is to understand the treatment use of luspatercept in adults diagnosed with lower-risk myelodysplastic syndromes

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary myelodysplastic syndromes (MDS) with lower-risk status as measured by the International Prognostic Scoring System (IPSS) or the Revised International Prognostic Scoring System (IPSS-R) at the time of diagnosis

  * IPSS risk level: low, intermediate-1 (level-1 risk)
  * IPSS-R risk level: very low, low, intermediate
* Initiated luspatercept for treatment of Lower-Risk (LR)-MDS after the initial availability in each country of interest

  * US: after April 2020
  * Germany: after June 2020
  * Spain: after June 2020
  * France: after June 202
  * Canada: after February 2021
* The participant has a potential follow-up of at least 6 months from the index date (except death)
* The participant is aged 18 years or older at the index date
* The participant has a complete medical record or history for at least 12 months before the index date (or up to the date of initial LR-MDS diagnosis if duration between initial diagnosis and index date is less than 12 months)

Exclusion Criteria:

* Received luspatercept as part of a clinical trial
* The participant has evidence of other malignant neoplasms prior to diagnosis of MDS, except disease free for ≥ 5 years at time of MDS diagnosis, basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, or incidental histologic finding of prostate cancer (stage T1a or T1b)
* The participant has a history of Acute Myeloid Leukemia prior to MDS diagnosis
* The participant has participated in clinical trials for specific treatments related to treatment of MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults diagnosed with lower-risk myelodysplastic syndromes (LR-MDS) who have been initiated luspatercept treatment in US, Germany, Spain, France and Canada
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
Participant baseline clinical characteristics | Baseline
Participant treatment history | Baseline

SECONDARY OUTCOMES:
Number of participants receiving myelodysplastic syndromes (MDS) -directed treatment modalities | Up to 12 months
  MDS-directed treatment modalities include:
  * Therapies for treatment of anemia include
    * Erythropoietin-stimulating agents (ESAs)
    * Granulocyte-colony stimulating factors (G-CSFs
    * Immunosuppressant/Immunomodulatory agents
    * Hypomethylating agents
    * Erythroid maturation agent
    * Other MDS-directed therapies
  * Other supportive care therapies
    * Antibiotic therapy
    * Iron chelation therapy
    * Nutritional support
Systemic therapy agent or combination of agents received by participants | Up to 12 months
Treating clinicians' rationale for prescribing treatment(s) | Up to 12 months
Time to treatment discontinuation | Up to 12 months
Duration of treatment | Up to 12 months
Reason(s) for treatment discontinuation | Up to 12 months
Treatment dosing characteristics | Up to 12 months
  Dosage characteristics includes:
  * Daily dose at treatment initiation
  * Dosing frequency
  * Dose modifications
  * Reason(s) for dose modification
  * Dose and dosing frequency at treatment discontinuation
Sequence of treatments prescribed to participants | Up to 12 months
Number and proportion of participants who received stem-cell transplant | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- RTI Health Solutions, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts